CLINICAL TRIAL: NCT06951269
Title: The Effect of Music Therapy on Pain Levels in Neonates With Hypoxic-ischemic Encephalopathy During Hypothermia: a Randomized Pilot and Feasibility Study
Brief Title: Music Therapy During Hypothermia in the NICU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Santa Fe de Bogota (Other)
Responsible Party: Principal Investigator, Mark Ettenberger, Principal Investigator, Music Therapy Service FSFB, Fundación Santa Fe de Bogota
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MTHYPOTHERMIA01
Record Dates: First submitted 2025-04-16; First posted 2025-04-30 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Music Therapy; Pain; Allodynia; Neonates; NICU; Hypothermia Neonatal
MeSH Terms: conditions — Pain; Hyperalgesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Main outcome measure will be evaluated through video analysis. The camera will be focused on the infant without the music therapist being in the frame. The sound will be muted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music therapy condition (Experimental): Live entrained music therapy
  Interventions: Behavioral: Live entrained music therapy
- Control condition (No Intervention): Standard care only

INTERVENTIONS:
Behavioral: Live entrained music therapy — This study will use live, improvised, entrainment-based music. The music will be applied to synchronize with the newborns' breathing patterns, adapting the tempo to the breathing rate, with characteristics that seek to induce a state of relaxation in the patient: moderate volume (below 65 dB; this measure will be validated using the ambient noise indicator of the neonatal intensive care unit), simple harmonic sequences (tonic-subdominant-dominant), melodies that avoid large intervals (beyond a third), medium registers, and a stable pulse. Once the music therapist synchronizes the pulse of the music with the newborn's breathing, the music will be gradually become slower (approximately 10-15%), the volume will be adjusted, and the complexity of the music will be reduced until the patient can transition to a state of greater relaxation. The music therapy session will last 10 minutes, after which the music therapist will leave the room.
  Arms: Music therapy condition

SUMMARY:
Background: Hypoxic-ischemic encephalopathy (HIE) is a neurological condition caused by poor oxygenation during the peripartum period. The main strategy to mitigate neurological damage is hypothermic therapy (HT), whose effectiveness-among other factors-depends on adequate pain management. Considering the prevalence of allodynia in this group of patients, routine nursing procedures can become sources of additional stress and pain. Music therapy is used in this population to promote self-regulation and relaxation, and may therefore help reduce pain levels after routine nursing procedures.

Research question: What is the effect of an entrainment-based live music therapy intervention on pain levels in newborns with hypoxic-ischemic encephalopathy undergoing hypothermic therapy after routine nursing procedures? Methodology: A randomized, crossover pilot and feasibility study. Participants will be 22 newborns admitted to the Neonatal Intensive Care Unit (NICU) of the University Hospital Fundación Santa Fe de Bogotá. Participants will receive standard care plus a 15-minute live music therapy session after a routine nursing procedure, or standard care alone. The primary outcome is the Premature Infant Pain Profile-Revised (PIPP-R) scale, which will be assessed through video recordings. Secondary outcomes are vital signs, heart rate variability, and electroencephalography (EEG) recordings.

Expected outcomes: Through this study, the aim is to improve the comfort and well-being of patients with HIE during TH. In addition, the safety and feasibility of music therapy in this population will be evaluated, seeking to contribute to current knowledge about the mechanisms of music therapy.

ELIGIBILITY:
Inclusion Criteria:

- Neonates diagnosed with neonatal hypoxic ischemic encephalopathy who have undergone hypothermic therapy as part of their medical treatment.

Exclusion Criteria:

* Newborns with a gestational age of less than 35 weeks and a birth weight of less than 1800 grams.
* Newborns in palliative care or with congenital anomalies with a poor prognosis will also be excluded, as will those with preexisting neurological or genetic conditions.
* Furthermore, newborns with a history of serious medical complications that may influence participation in the study, such as pulmonary hypertension or secondary seizure syndrome, will be considered ineligible.
* Finally, patients with an N-PASS score of less than -2 will be excluded.

Ages: 35 Weeks to 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Premature Infant Pain Profile - Revised (PIPP-R) | From start of the conditions to the end of the conditions, for about 30 minutes
  The Premature Infant Pain Profile - Revised (PIPP-R) is a 10-item pain score used to assess pain in term and preterm infants. It consists of three indicators: physiological, e.g., heart rate and oxygen saturation; behavioral, e.g., facial expression; and contextual, e.g., gestational age. In the present study, for the behavioural part of the the PIPP-R we will use video recordings of the infant's face. Two raters will identify facial expressions associated with pain through one-minute video segments. The audio will be removed from the video, and measures will be taken to ensure that the music therapist does not appear in the recording, thus keeping the raters masked to the type of intervention.

SECONDARY OUTCOMES:
Heart rate | From start of the conditions to the end of the conditions, for about 30 minutes.
  Heart rate will be measured in beats per minute (BPM) and will be recorded continuously from 5 minutes before the routine nursing procedure, during the routine nursing procedure, during the music therapy intervention or the control condition, and up to 5 minutes after the intervention.
Heart rate variability | From start of the conditions to the end of the conditions, for about 30 minutes.
  Telemetry recordings will be used to obtain electrocardiographic time series. This measurement provides an estimate of sympathetic and vagal tone, which has been linked to the outcome of infants with HIE during HT.
EEG - Electroencelography | From start of the conditions to the end of the conditions, for about 30 minutes.
  Video telemetry recordings will be visually analyzed by the neurologist for patterns of seizure and abnormal activity; excessive discontinuities in the tracing, low voltage, or suppression of normal burst activity will be sought. These indicators correlate with the prognosis of the neonate with HIE during TH, the preservation of brain tissue, and the safety of the MT intervention.
Oxygen saturation | From start of the conditions to the end of the conditions, for about 30 minutes.
  Oxygen saturation will be measured in percentage (%) and will be recorded continuously from 5 minutes before the routine nursing procedure, during the routine nursing procedure, during the music therapy intervention or the control condition, and up to 5 minutes after the intervention.
Respiratory Rate | From start of the conditions to the end of the conditions, for about 30 minutes.
  Respiratory rate will be measured in numbers of respirations per minute and will be recorded continuously from 5 minutes before the routine nursing procedure, during the routine nursing procedure, during the music therapy intervention or the control condition, and up to 5 minutes after the intervention.

OTHER OUTCOMES:
Viability and safety measures | From start of the conditions to the end of the conditions, for about 30 minutes.
  Number of events indicating hemodynamic instability or a negative change in vital signs during music therapy interventions and number of epileptic events during music therapy interventions. If music therapy sessions are discontinued in more than three patients, the study will be discontinued.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Fundación Santa Fe de Bogotá, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon request
Supporting Information: Study Protocol
Time Frame: data will be available after publication of the results